CLINICAL TRIAL: NCT04152200
Title: ILLUMINATE-C: A Single Arm Study to Evaluate Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Lumasiran in Patients With Advanced Primary Hyperoxaluria Type 1 (PH1)
Brief Title: A Study to Evaluate Lumasiran in Patients With Advanced Primary Hyperoxaluria Type 1
Acronym: ILLUMINATE-C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-GO1-005; 2019-001346-17 (EudraCT Number); 2023-503382-29-00 (EU CTIS Number)
Expanded Access: NCT04125472 (Approved for marketing)
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Results first posted 2022-07-12 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Primary Hyperoxaluria Type 1; Primary Hyperoxaluria
Keywords: PH1; Primary Hyperoxaluria; Hyperoxaluria; RNAi Therapeutic; siRNA; AGT; Systemic Oxalosis
MeSH Terms: conditions — Primary hyperoxaluria type 1; Hyperoxaluria, Primary; Hyperoxaluria | interventions — lumasiran

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lumasiran (Experimental): All patients will receive open-label lumasiran.
  Interventions: Drug: Lumasiran

INTERVENTIONS:
Drug: Lumasiran — Lumasiran will be administered by subcutaneous (SC) injection.
  Other Names: ALN-GO1; OXLUMO

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, pharmacokinetics (PK), and pharmacodynamics (PD) of lumasiran in patients with Advanced Primary Hyperoxaluria Type 1 (PH1).

ELIGIBILITY:
Inclusion Criteria:

* Has documented diagnosis of primary hyperoxaluria type 1 (PH1)
* Estimated glomerular filtration rate (eGFR) ≤45 mL/min/1.73 m^2 for patients ≥12 months of age (<12 months of age, must have serum creatinine considered elevated for age)
* Meets plasma oxalate level requirements
* If taking Vitamin B6 (pyridoxine), must have been on stable regimen for at least 90 days
* If on dialysis, may be on hemodialysis therapy only and must have been on a stable regimen for at least 4 weeks

Exclusion Criteria:

* Hemodialysis/peritoneal dialysis combination therapy or peritoneal dialysis alone
* Diagnosis of conditions other than PH1 contributing to renal insufficiency
* History of liver transplant
* History of kidney transplant and currently receiving immunosuppressants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2025-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (14):
- United States (2):
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, Houston, Texas
- Clinical Trial Site, Garran, Australia
- Clinical Trial Site, Brussels, Belgium
- France (2):
  - Clinical Trial Site, Bron
  - Clinical Trial Site, Lyon
- Israel (2):
  - Clinical Trial Site, Haifa
  - Clinical Trial Site, Nahariya
- Clinical Trial Site, Rome, Italy
- Clinical Trial Site, Irbid, Jordan
- Clinical Trial Site, Beirut, Lebanon
- Clinical Trial Site, Amsterdam, Netherlands
- Clinical Trial Site, Yenimahalle, Turkey (Türkiye)
- Clinical Trial Site, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Requests for access to data can be submitted via the website www.vivli.org.

REFERENCES:
- [Derived] Michael M, Groothoff JW, Shasha-Lavsky H, Lieske JC, Frishberg Y, Simkova E, Sellier-Leclerc AL, Devresse A, Guebre-Egziabher F, Bakkaloglu SA, Mourani C, Saqan R, Singer R, Willey R, Habtemariam B, Gansner JM, Bhan I, McGregor T, Magen D. Lumasiran for Advanced Primary Hyperoxaluria Type 1: Phase 3 ILLUMINATE-C Trial. Am J Kidney Dis. 2023 Feb;81(2):145-155.e1. doi: 10.1053/j.ajkd.2022.05.012. Epub 2022 Jul 14. PMID 35843439

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with advanced primary hyperoxaluria type 1 (PH1) were enrolled at thirteen sites in Australia, Belgium, France, Israel, Jordan, Lebanon, the Netherlands, Turkey, the United Arab Emirates and the United States.
Groups:
- Cohort A: Lumasiran: Patients not on dialysis received open-label lumasiran based on weight. Patients weighing <10 kg received loading doses of lumasiran subcutaneous (SC) injection 6.0 mg/kg monthly for 3 months, followed by maintenance doses of lumasiran SC injection 3.0 mg/kg monthly during the 6-month primary analysis period and monthly during the 54-month extension period. Patients in maintenance dosing who transitioned from <10 kg to ≥10 kg continued to receive monthly doses at 3.0 mg/kg until the next visit that coincided with a dose for patients weighing ≥10 kg. Thereafter, patients followed every-3-months dosing until the end of the study. Patients weighing ≥10 to <20 kg received loading doses of lumasiran SC injection 6.0 mg/kg monthly for 3 months, followed by maintenance doses of lumasiran SC injection 6.0 mg/kg at Months 3 and 6 in the 6-month primary analysis period and every three months during the 54-month extension period. Patients weighing ≥20 kg received loading doses of lumasiran SC injection 3.0 mg/kg monthly for 3 months, followed by maintenance doses of lumasiran SC injection 3.0 mg/kg at Months 3 and 6 in the 6-month primary analysis period and every three months during the 54-month extension period. Patients with weight increases crossing the threshold for the next weight-based dosing category (<10 kg to ≥10 kg or <20 kg to ≥20 kg) followed the new dosing regimen for the remainder of the study or until the next dosing category threshold was reached.
- Cohort B: Lumasiran: Patients on dialysis received open-label lumasiran based on weight. Patients weighing <10 kg received loading doses of lumasiran subcutaneous (SC) injection 6.0 mg/kg monthly for 3 months, followed by maintenance doses of lumasiran SC injection 3.0 mg/kg monthly during the 6-month primary analysis period and monthly during the 54-month extension period. Patients in maintenance dosing who transitioned from <10 kg to ≥10 kg continued to receive monthly doses at 3.0 mg/kg until the next visit that coincided with a dose for patients weighing ≥10 kg. Thereafter, patients followed every-3-months dosing until the end of the study. Patients weighing ≥10 to <20 kg received loading doses of lumasiran SC injection 6.0 mg/kg monthly for 3 months, followed by maintenance doses of lumasiran SC injection 6.0 mg/kg at Months 3 and 6 in the 6-month primary analysis period and every three months during the 54-month extension period. Patients weighing ≥20 kg received loading doses of lumasiran SC injection 3.0 mg/kg monthly for 3 months, followed by maintenance doses of lumasiran SC injection 3.0 mg/kg at Months 3 and 6 in the 6-month primary analysis period and every three months during the 54-month extension period. Patients with weight increases crossing the threshold for the next weight-based dosing category (<10 kg to ≥10 kg or <20 kg to ≥20 kg) followed the new dosing regimen for the remainder of the study or until the next dosing category threshold was reached.
Period: Primary Analysis Period
Arm/Group | Cohort A: Lumasiran | Cohort B: Lumasiran
Started | 6 | 15
Completed | 6 | 15
Not Completed | 0 | 0
Period: Long-term Extension Period
Arm/Group | Cohort A: Lumasiran | Cohort B: Lumasiran
Started | 6 | 15
Completed | 0 | 0
Not Completed | 6 | 15
Not completed — Entered Long-term Extension Period after completion of the Primary Analysis Period | 6 | 15

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS): All patients who received any amount of lumasiran during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Lumasiran | Cohort B: Lumasiran | Total
Number analyzed (Participants) | 6 | 15 | 21
Age, Continuous [Median (Full Range); unit: years] | 9.0 [0 to 40] | 6.0 [1 to 59] | 8.0 [0 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 3 | 9 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 3 | 4
  White | 4 | 12 | 16
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 14 | 20
Plasma Oxalate [Mean (Standard Deviation); unit: μmol/L] — For Cohort A, the baseline was defined as the mean of all plasma oxalate samples collected prior to the first dose of lumasiran; for Cohort B the baseline was defined as the mean of the last 4 pre-dialysis plasma oxalate samples collected prior to the first dose of lumasiran. In Cohort B, only pre-dialysis samples were utilized.
  μmol/L | 64.73 (41.30) | 108.35 (29.53) | 95.89 (38.01)

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Percent Change in Plasma Oxalate From Baseline to Month 6
Description: Percent change in plasma oxalate (umol/L) was estimated by an average percent change from baseline across Months 3 through 6. A negative change from Baseline indicates a favorable outcome. For Cohort A, the baseline was defined as the mean of all plasma oxalate level values collected prior to the first dose of lumasiran.
Time Frame: Baseline to Month 6
Population: Full Analysis Set (FAS): All patients who received any amount of lumasiran and had at least 1 evaluable plasma oxalate value (pre-dialysis in Cohort B) at baseline and at least 1 evaluable plasma oxalate value from assessment(s) at Month 3 through Month 6.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Cohort A: Lumasiran
Number analyzed (Participants) | 6
percent change | -33.33 (17.63)
Statistical Analysis 1: Comparison: Cohort A: Lumasiran; Restricted maximum likelihood (REML) based Mixed Model Repeated Measures (MMRM) was used to test against the null hypothesis of mean change from baseline outcome being equal to 0. The model includes scheduled visits and baseline plasma oxalate (μmol/L) as fixed effects and patient as a random factor. Autoregressive (1) was used to model the within-patient variability; Test type: Other — Not applied; Mixed model repeated measures (MMRM); Least Squares (LS) Mean = -33.33, 95% CI 2-sided [-81.82 to 15.16], Standard Error of Mean 17.63

2. Primary Outcome: Cohort B: Percent Change in Pre-dialysis Plasma Oxalate From Baseline to Month 6
Description: Percent change in plasma oxalate (umol/L) was estimated by an average percent change from baseline across Months 3 through 6. A negative change from Baseline indicates a favorable outcome. For Cohort B, the baseline is defined as the mean of the last four pre-dialysis plasma oxalate samples collected prior to the first dose of lumasiran. In Cohort B, only pre-dialysis samples are utilized.
Time Frame: Baseline to Month 6
Population: FAS: All patients who received any amount of lumasiran and had at least 1 evaluable plasma oxalate value (pre-dialysis in Cohort B) at baseline and at least 1 evaluable plasma oxalate value from assessment(s) at Month 3 through Month 6.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Cohort B: Lumasiran
Number analyzed (Participants) | 15
percent change | -42.43 (3.95)
Statistical Analysis 1: Comparison: Cohort B: Lumasiran; REML based Mixed Model Repeated Measures MMRM was used to test against the null hypothesis of mean change from baseline outcome being equal to 0. The model includes scheduled visits and baseline plasma oxalate (μmol/L) as fixed effects and patient as a random factor. Autoregressive (1) was used to model the within-patient variability; Test type: Other — Not applied; MMRM; Least Squares (LS) Mean = -42.43, 95% CI 2-sided [-50.71 to -34.15], Standard Error of Mean 3.95

3. Secondary Outcome: Cohort B: Percent Change in Plasma Oxalate Area Under the Curve From 0-24 Hours [AUC(0-24)] Between Dialysis Sessions From Baseline to Month 6
Description: Percent change in plasma oxalate AUC(0-24) was estimated by an average percent change from baseline across Months 3 through 6. A negative change from Baseline indicates a favorable outcome. Baseline was defined as the mean value of all valid AUC (μmol/L/24h) profiles being computed prior to the first dose of lumasiran.
Time Frame: Baseline to Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Cohort B: Lumasiran
Number analyzed (Participants) | 15
percent change | -41.4 (4.4)

4. Secondary Outcome: Absolute Change in Plasma Oxalate From Baseline to Month 6
Description: Absolute change in plasma oxalate was estimated by an average absolute change from baseline across Months 3 through 6. A negative change from Baseline indicates a favorable outcome. For Cohort A, the baseline was defined as the mean of all plasma oxalate level values collected prior to the first dose of lumasiran; for Cohort B, the baseline was defined as the mean of the last 4 pre-dialysis plasma oxalate level values collected prior to the first dose of lumasiran. In Cohort B patients, the plasma oxalate baseline was similarly defined except that the values obtained from the plasma oxalate profile assessment visits only included the pre-dialysis sample collected per visit.
Time Frame: Baseline to Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Cohort A: Lumasiran | Cohort B: Lumasiran
Number analyzed (Participants) | 6 | 15
μmol/L | -35.28 (7.40) | -48.33 (3.63)

5. Secondary Outcome: Cohort A: Absolute Change in 24-hour Urinary Oxalate Excretion Corrected for Body Surface Area (BSA) From Baseline to Month 6
Description: Absolute change in 24-hour urinary oxalate excretion corrected for BSA was estimated by an average absolute change from baseline across Months 3 through 6. Only valid urine samples without any non-protocol-related issues were included in the analysis. A negative change from Baseline indicates a favorable outcome. Baseline is defined as the median of all valid 24-hr urine assessments collected prior to the first dose date/time of lumasiran without any non-protocol-related sample issues.
Time Frame: Baseline to Month 6
Population: FAS: All patients who received any amount of lumasiran (with data available for analysis) and had at least 1 evaluable plasma oxalate value (pre-dialysis in Cohort B) at baseline and at least 1 evaluable plasma oxalate value from assessment(s) at Month 3 through Month 6. No analyses were performed for patients in Cohort B that were anuric (ie, patients able to continue to produce urine ≥100 mL per day).
Measure: Least Squares Mean (Standard Error); unit: mmol/24hr/1.73m^2
Arm/Group | Cohort A: Lumasiran
Number analyzed (Participants) | 5
mmol/24hr/1.73m^2 | -0.533 (0.111)

6. Secondary Outcome: Cohort A: Percent Change in 24-hour Urinary Oxalate Excretion Corrected for Body Surface Area (BSA) From Baseline to Month 6
Description: Percent change in 24-hour urinary oxalate excretion corrected for BSA was estimated by an average percent change from baseline across Months 3 through 6. Only valid urine samples without any non-protocol-related issues were included in the analysis. A negative change from Baseline indicates a favorable outcome. Baseline is defined as the mean of all assessments prior to the first dose date/time of lumasiran.
Time Frame: Baseline to Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Cohort A: Lumasiran
Number analyzed (Participants) | 5
percent change | -10.557 (6.811)

7. Secondary Outcome: Cohort A: Absolute Change in Spot Urinary Oxalate:Creatinine Ratio From Baseline to Month 6
Description: Absolute change in spot urinary oxalate:creatinine ratio was estimated by an average absolute change from baseline across Months 3 through 6. A negative change from Baseline indicates a favorable outcome. Baseline was defined as the mean of all assessments prior to the first dose date/time of lumasiran.
Time Frame: Baseline to Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Cohort A: Lumasiran
Number analyzed (Participants) | 6
ratio | -0.1879 (0.0160)

8. Secondary Outcome: Cohort A: Percent Change in Spot Urinary Oxalate:Creatinine Ratio From Baseline to Month 6
Description: Percent change in spot urinary oxalate:creatinine ratio was estimated by an average percent change from baseline across Months 3 through 6. A negative change from Baseline indicates a favorable outcome. Baseline was defined as the mean of all assessments prior to the first dose date/time of lumasiran.
Time Frame: Baseline to Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Cohort A: Lumasiran
Number analyzed (Participants) | 6
percent change | -39.5136 (9.4294)

9. Secondary Outcome: Change in Quality of Life As Assessed by Pediatric Quality of Life Inventory (PedsQL) Total Score From Baseline to Month 6 in Patients >=2 to 18 Years of Age at Time of Informed Consent
Description: Peds-QL is a modular approach to measuring quality of life (QOL) in healthy children and adolescents and those with acute and chronic health conditions. The PedsQL Generic Core Scales contain 23 items designed to measure core domains of health (physical, emotional, and social functioning) and role (school functioning). Scores are summarized as Total Scale Score, Physical Health Summary Score, and Psychosocial Health Summary Score. The Total Scale Score will be reported for this study. The PedsQL will be completed by patients (or caregivers, as appropriate) who are ≥2 to <18 years of age at the time of consent. Total score range: 0 - 100, with higher scores indicating better health-related quality of life (HRQoL). Baseline is defined as last non-missing value collected prior to the first dose of lumasiran.
Time Frame: Baseline to Month 6
Population: Participants from the FAS who were ≥2 to <18 years of age at the time of consent with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A: Lumasiran | Cohort B: Lumasiran
Number analyzed (Participants) | 2 | 5
score on a scale | -23.91 (9.22) | 0.10 (8.52)

10. Secondary Outcome: Change in Quality of Life As Assessed by Kidney Disease and Quality of Life (KDQOL) Scores From Baseline to Month 6 in Patients ≥18 Years of Age at Time of Informed Consent
Description: The KDQOL questionnaire is used to assess 3 core domains of kidney disease including: burden, symptoms/problems, and effects of kidney disease on daily life. The KDQOL subscales (Burden of Kidney Disease, Effect of Kidney Disease on Daily Life, and Symptoms and Problems of Kidney Disease), and the accompanying Short Form-12 (SF-12) Physical Component Summary and Mental Component Summary will be assessed for this study. These will be completed by patients who are ≥18 years of age at the time of consent. Score range (per domain): 0 - 100; higher scores indicate better HRQoL. Baseline is defined as last non-missing value collected prior to the first dose of lumasiran.
Time Frame: Baseline to Month 6
Population: Participants from the FAS who were ≥18 years of age at the time of consent.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A: Lumasiran | Cohort B: Lumasiran
Number analyzed (Participants) | 2 | 4
score on a scale
  SF-12 Physical Component Score | -1.56 (1.19) | -2.06 (6.59)
  SF-12 Mental Component Score | -3.88 (4.45) | 1.58 (9.61)
  Symptoms/Problems of Kidney Disease | -13.64 (6.43) | -5.73 (7.49)
  Effects of Kidney Disease | -15.63 (22.10) | -10.16 (14.96)
  Burden of Kidney Disease | -3.13 (4.42) | -4.69 (16.44)

11. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Lumasiran
Description: Cmax is the highest concentration of lumasiran in the plasma after a dose is given.
Time Frame: Day 1; Month 6
Population: Pharmacokinetic (PK) Analysis Set: All patients who received any amount of lumasiran, have at least 1 postdose blood sample for PK parameters, and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- All Lumasiran: All patients from Cohorts A and B.
Arm/Group | Cohort A: Lumasiran | Cohort B: Lumasiran | All Lumasiran
Number analyzed (Participants) | 6 | 15 | 21
ng/mL
  Day 1 | 1019.9 (61.6) | 1820.5 (113.2) | 1542.8 (103.7)
  Month 6 | 1038.2 (36.9) | 1289.3 (106.0) | 1211.9 (87.6)

12. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Lumasiran
Description: Tmax is the time it takes for lumasiran to reach the maximum concentration (Cmax) after administration.
Time Frame: Day 1; Month 6
Population: PK Analysis Set: All patients who received any amount of lumasiran, have at least 1 postdose blood sample for PK parameters, and have evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A: Lumasiran | Cohort B: Lumasiran | All Lumasiran
Number analyzed (Participants) | 6 | 15 | 21
hours
  Day 1 | 3.8083 [1.767 to 11.533] | 4.0000 [1.717 to 12.000] | 4.0000 [1.717 to 12.000]
  Month 6 | 3.9083 [1.983 to 7.617] | 4.0167 [1.967 to 12.000] | 4.0000 [1.967 to 12.000]

13. Secondary Outcome: Elimination Half-life (t½β) of Lumasiran
Description: t½β is the time it takes for the concentration of the drug in the plasma to be reduced by 50%.
Time Frame: Day 1; Month 6
Population: PK Analysis Set: All patients who received any amount of lumasiran, have at least 1 postdose blood sample for PK parameters, and have evaluable PK data at the given timepoint.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A: Lumasiran | Cohort B: Lumasiran | All Lumasiran
Number analyzed (Participants) | 6 | 15 | 21
hours
  Day 1: number analyzed (Participants) | 3 | 8 | 11
  Day 1 | 9.0246 [3.364 to 10.593] | 3.6670 [1.127 to 7.793] | 3.8302 [1.127 to 10.593]
  Month 6: number analyzed (Participants) | 3 | 4 | 7
  Month 6 | 8.1069 [2.420 to 10.796] | 4.5131 [1.388 to 7.354] | 5.7484 [1.388 to 10.796]

14. Secondary Outcome: Area Under the Concentration-time Curve From 0 to 24 Hours [AUC(0-24)] for Lumasiran
Description: AUC(0-24) is the area under the plasma concentration-time curve over the last 24-h dosing interval.
Time Frame: Day 1; Month 6
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort A: Lumasiran | Cohort B: Lumasiran | All Lumasiran
Number analyzed (Participants) | 6 | 15 | 21
h*ng/mL
  Day 1: number analyzed (Participants) | 6 | 7 | 13
  Day 1 | 13156.8031 (64.6) | 13170.3716 (35.6) | 13164.1075 (47.7)
  Month 6: number analyzed (Participants) | 5 | 4 | 9
  Month 6 | 11417.0267 (33.5) | 20647.6317 (61.6) | 14856.4905 (55.9)

15. Secondary Outcome: Apparent Clearance (CL/F) of Lumasiran
Description: CL/F is the rate at which lumasiran is eliminated from the body.
Time Frame: Day 1; Month 6
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour (L/h)
Arm/Group | Cohort A: Lumasiran | Cohort B: Lumasiran | All Lumasiran
Number analyzed (Participants) | 6 | 15 | 21
Liters/hour (L/h)
  Day 1: number analyzed (Participants) | 3 | 8 | 11
  Day 1 | 7.8440 (105.5) | 5.1003 (77.7) | 5.7356 (82.6)
  Month 6: number analyzed (Participants) | 3 | 4 | 7
  Month 6 | 4.8496 (112.8) | 6.8556 (44.8) | 5.9104 (70.1)

16. Secondary Outcome: Apparent Volume of Distribution (V/F) of Lumasiran
Description: V/F is the propensity of lumasiran to either remain in the plasma or redistribute to other tissues.
Time Frame: Day 1; Month 6
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Cohort A: Lumasiran | Cohort B: Lumasiran | All Lumasiran
Number analyzed (Participants) | 6 | 15 | 21
Liters (L)
  Day 1: number analyzed (Participants) | 3 | 8 | 11
  Day 1 | 77.5329 (91.1) | 25.7429 (196.4) | 34.7734 (185.7)
  Month 6: number analyzed (Participants) | 3 | 4 | 7
  Month 6 | 41.7081 (229.3) | 36.8305 (166.9) | 38.8468 (161.3)

17. Secondary Outcome: Percent Change in Plasma Oxalate Area Under the Curve From 0-24 Hours [AUC(0-24)] Between Dialysis Sessions From Baseline to Month 60
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

18. Secondary Outcome: Absolute Change in Plasma Oxalate From Baseline to Month 60
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

19. Secondary Outcome: Absolute Change in 24-hour Urinary Oxalate Excretion Corrected for Body Surface Area (BSA) From Baseline to Month 60
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

20. Secondary Outcome: Percent Change in 24-hour Urinary Oxalate Excretion Corrected for Body Surface Area (BSA) From Baseline to Month 60
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

21. Secondary Outcome: Absolute Change in Spot Urinary Oxalate:Creatinine Ratio From Baseline to Month 60
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

22. Secondary Outcome: Percent Change in Spot Urinary Oxalate:Creatinine Ratio From Baseline to Month 60
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

23. Secondary Outcome: Change in Quality of Life As Assessed by Pediatric Quality of Life Inventory (PedsQL) Total Score From Baseline to Month 60 in Patients >=2 to 18 Years of Age at Time of Informed Consent
Description: as for outcome 9
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

24. Secondary Outcome: Change in Quality of Life As Assessed by Kidney Disease and Quality of Life (KDQOL) Scores From Baseline to Month 60 in Patients ≥18 Years of Age at Time of Informed Consent
Description: as for outcome 10
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

25. Secondary Outcome: Percent Change in Plasma Oxalate From Baseline to End of Study
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

26. Secondary Outcome: Change in Nephrocalcinosis From Baseline to End of Study
Description: Nephrocalcinosis will be assessed by renal ultrasound.
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

27. Secondary Outcome: Change in Frequency of Dialysis From Baseline to End of Study
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

28. Secondary Outcome: Change in Mode of Dialysis From Baseline to End of Study
Description: Modes of dialysis are defined as hemodialysis and peritoneal dialysis.
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

29. Secondary Outcome: Change in Frequency of Renal Stone Events From Baseline to End of Study
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

30. Secondary Outcome: Change in Renal Function Assessed by Estimated Glomerular Filtration Rate (eGFR) From Baseline to End of Study
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

31. Secondary Outcome: Change in Measures of Systemic Oxalosis From Baseline to End of Study
Description: Systemic oxalosis will be assessed in cardiac, skeletal, ophthalmologic, and dermatologic systems.
Time Frame: Baseline to Month 60
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (AEs) are reported from the administration of the first dose of study drug up to approximately 6 months. Serious adverse events (SAEs) are reported from the time when the informed consent is signed up to approximately 6 months.
Arm/Group | Cohort A: Lumasiran | Cohort B: Lumasiran
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/6 | 8/15
Other Adverse Events (participants affected / at risk) | 5/6 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Lumasiran (N=6) | Cohort B: Lumasiran (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Catheter site swelling (General disorders) | 0 | 1
Device related thrombosis (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Device related infection (Infections and infestations) | 0 | 2
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Skin scar contracture (Injury, poisoning and procedural complications) | 0 | 1
General physical condition abnormal (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 0 | 1
Dialysis device insertion (Surgical and medical procedures) | 0 | 1
Renal and liver transplant (Surgical and medical procedures) | 0 | 1
Renal transplant (Surgical and medical procedures) | 0 | 2
Haemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Lumasiran (N=6) | Cohort B: Lumasiran (N=15)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Gastritis (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Injection site reaction (General disorders) | 1 | 4
Pyrexia (General disorders) | 1 | 6
Swelling (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Candida nappy rash (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 2
Ear infection (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Roseola (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood phosphorus increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 2
Staphylococcus test positive (Investigations) | 0 | 1
Carnitine deficiency (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Thrombosis in device (Product Issues) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dialysis hypotension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. Copy of disclosure is provided to Sponsor at least 60 days before submission for publication or date of disclosure
2. Confidential information is deleted if requested by Sponsor
3. If a Discovery is disclosed, defer publication or disclosure for 60 days from time Sponsor notifies them of its wish to file a patent application on such Discovery
4. Site/Investigator will not disclose or publish results until results from all sites have been received and analyzed by Sponsor

DOCUMENTS (2):
  • Study Protocol (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT04152200/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT04152200/SAP_001.pdf